CLINICAL TRIAL: NCT05176730
Title: Effects of Mindfulness Meditation on Trait Mindfulness, Perceived Stress, Emotion Regulation, and Quality of Life in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Mindfulness Meditation For Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 731-2020
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Diseases; Hemodialysis Complication
Keywords: Hemodialysis; Stress; Emotion regulation; Mindfulness meditation; Quality of life; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Emotional Regulation | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A repeated-measure, two-group, randomized design
Who Masked: Outcomes Assessor
Masking Description: The data were collected by three research assistants with at least 10 years nursing experiences who were not involved in any other parts of the study.
  Also, the participants were randomly assigned equally to the study groups using a computerized random numbers procedure carried out by a research assistant who was not involved in any other parts of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with hemodialysis receiving mindfulness meditation (Experimental): The ABC standardized version of mindfulness meditation was used. The experimental group received 30-minute mindfulness meditation sessions 3 times a week for 5 weeks (450 minutes). An additional two-hour educational workshop about the rationale and procedures of intervention was provided before the actual training sessions. To ensure the consistent delivery of the intervention, the researcher recorded the intervention instructions in Arabic based on the intervention protocol and sent the audio-recorded instructions to the participants via WhatsApp or email. The audio-recorded intervention contents were validated by two psychologists and experts in meditation. The recorded intervention instructions were accessed by the participants during the sessions using their cell phones and headsets, as recommended. This method allowed for up to 3-5 participants to listen to the instructions and perform the intervention simultaneously.
  Interventions: Behavioral: Mindfulness meditation
- Control group (No Intervention): The participants in the control group were instructed to sit with their eyes closed and relaxed for 30 minutes 3 times a week for 5 weeks during hemodialysis sessions to control for the nonspecific effects of social interaction and environment. The timings of the control group sessions were similar to those of the experimental group, whereby if a given experimental group intervention lasted for 30 minutes, the control group participants would be asked to sit with their eyes closed and relax for 30 minutes also.

INTERVENTIONS:
Behavioral: Mindfulness meditation — Similar to the information included in arm/group descriptions
  Arms: Patients with hemodialysis receiving mindfulness meditation

SUMMARY:
Objective: This study aimed to examine the effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in end-stage renal disease patients undergoing hemodialysis.

Method: An experimental repeated measures design was used among a sample of 74 end-stage renal disease patients undergoing hemodialysis at a dialysis center at Jahra hospital, Kuwait. The patients were randomly assigned to the experimental (n=37) and control groups (n=37). The experimental group participated in 30-minute mindfulness meditation sessions (three sessions a week for five weeks) held during their hemodialysis sessions. The dependent variables of both groups were measured at baseline, middle of intervention, and end of intervention using the Mindful Attention Awareness Scale (MAAS), Perceived Stress Scale (PSS), Emotion Regulation Questionnaire (ERQ), and Kidney Disease Quality of Life (KDQOL-36) questionnaire.

DETAILED DESCRIPTION:
Introduction

End-stage renal disease (ESRD) has been reported to be a major cause of disability and increased mortality worldwide. In patients with ESRD, hemodialysis is a critically vital therapy that prolongs survival and improves quality of life through the excretion or removal of poisonous metabolic waste from the human body. However, compliance with treatment has been found to be poor among ESRD patients. Such incompliance can be attributed to the different sources of stress associated with hemodialysis, including hemodialysis complications, time-consuming treatment schedules, restriction of dietary and fluid intake, and prescription of multiple medications. These sources of stress, in addition to the signs and symptoms of ESRD, result in diminished health-related quality of life, which is associated with increased risks of morbidity, mortality, and incompliance with hemodialysis therapy.

Despite the significant physical, emotional, and social burdens of stress, stress-reduction strategies have been inadequately used in patients undergoing hemodialysis. This may be contributed to the small-scale studies on psychotherapies with variable and holistic outcomes and the limited availability of evidenced-based coping interventions that are significantly supported. Mind-body therapies, which comprise a variety of techniques that increase the capacity of the mind to influence the functions of the body using emotional strategies, have gained increasing popularity worldwide in recent years. Evidence shows that mind-body therapies are affordable, easily-practiced, and safe, and that they improve perceived stress, health-related outcomes, and quality of life among various community-dwelling and clinical populations. One of the most popular mind-body therapies in the literature is mindfulness meditation, which has been found to be a feasible, beneficial, and well-tolerated therapy in hemodialysis patients.

It is theoretically claimed that mindfulness meditation can positively impact perceived stress, known also as stress appraisal, and quality of life through the improvement of trait mindfulness and emotion regulation. Hemodialysis is appraised as an uncontrollable, threatening situation, since hemodialysis patients must undergo hemodialysis for their entire lives for survival. Therefore, hemodialysis is not a cure for terminal renal diseases but rather a maintenance therapy. It is claimed that repeated mindfulness-based practices cultivate and improve the natural mental capacity of mindfulness, called trait mindfulness. Trait mindfulness is described as the mental capacity to pay attention to, be aware of, and accept current experiences in a non-judgmental way. This developed mental capacity enables psychological distance through a process of decentered attention, through which one's attention (e.g., thoughts, emotions, and sensations) shifts from the contents of consciousness to the process of consciousness itself. In turn, this can help to stop initial automatic uncontrollable appraisals and broaden attention and awareness to include previously overlooked positive aspects of self, context, or events. Based on this new information, it becomes possible to flexibly select adaptive responses and to reappraise events as beneficial or meaningful (i.e., positive reappraisals). Trait mindfulness also enables individuals to acknowledge and accept their current experiences, even if these experiences are uncomfortable. In addition, trait mindfulness helps individuals to not engage in judgmental or negative thinking or avoidance of these experiences, resulting in less reactivity to stressful situations and increased quality of life.

Research supports these theoretical claims, whereby mindfulness meditation has been found to be highly effective for a variety of health outcomes in several psychiatric and medical illnesses. For patients undergoing hemodialysis specifically, studies have demonstrated that mindfulness meditation significantly improves trait mindfulness, stress symptoms, emotion regulation, and quality of life and general health. However, these studies have serious limitations that limit the validity and generalizability of their findings. For example, these studies generally used small samples, in addition to inconsistent intervention protocols in terms of the intervention contents and duration. Further, no study has examined the effectiveness of mindfulness-based interventions among patients undergoing hemodialysis in Kuwait. Therefore, the current study aimed to examine the effects of a mindfulness-based intervention on trait mindfulness, perceived stress, emotion regulation, and health-related quality of life in ESRD patients undergoing hemodialysis.

Theoretically, investigating the effects of mindfulness meditation on the selected variables may provide insight into the mechanisms through which mindfulness meditation impacts quality of life in hemodialysis patients. The current study findings may enrich the body of knowledge on mindfulness meditation and bridge the gap in the literature regarding the effects of mindfulness meditation on patients receiving hemodialysis. Practically, the findings of the present study may guide decision-makers in adopting mindfulness meditation in hospitals.

Methods

Design

This study used a repeated-measures, randomized, wait-list, control design and was conducted in the dialysis center at Jahra Hospital, Kuwait. Seventy-four ESRD patients undergoing hemodialysis were recruited using convenience sampling. Jahra Hospital is a governmental hospital with one of the biggest dialysis centers in Kuwait, with a female ward, male ward, and isolation ward. The center holds 70 dialysis machines/beds, with an average number of 30 patients managed per day.A research assistant, who was not involved in the recruitment or patient assessment processes, randomly assigned the participants to the intervention group (n=37) or the control group (n=37) using a simple 1:1 computer-generated sequence. The trial is reported in accordance with the CONSORT guideline.

Determination of the Sample Size

The required sample size was calculated using G-power version (3.1). Given a mixed-design (within groups and between groups) repeated measures ANOVA, power of 0.95, moderate effect size of 0.25, and α of .0125, the required sample size was 56 subjects. Taking into consideration a 60% attrition rate, the final total sample size was 89 patients.

Intervention

The experimental group received the Smith's version of mindfulness meditation, which is a standardized theory-based intervention found to be effective in improving stress and its related health problems. The Smith's version of mindfulness meditation comprises the following components:

1. Being mindful of breathing, which includes easily taking in a full, deep breath, filling the lungs, simply exhaling, and then breathing naturally. It also includes noticing and simply attending to the air as it flows in and out of the nose and moves deeper into the throat and lungs (5 minutes).
2. Being mindful of the body, which includes attending to how the body feels from head to toes and noticing any sensations that come and go. Upon noticing a sensation, the individual must gently note it, let it go, and continue attending to how the body feels (5 minutes).
3. Being mindful of thought, which includes attending to the mind as thoughts come and go. Whenever a thought or feeling comes to mind, the individual should just notice it, let it go, and continue attending to the mind repeatedly (5 minutes).
4. Being mindful of sounds, which includes attending to the sounds one hears, without thinking about them. The individual must gently notice the sound, let it go, and continuing waiting (5 minutes).
5. Being mindful of taste, which includes imagining a wonderful bowl of pieces of one's favorite fruit and simply attending to a taste sensation, without thought, analysis, or effort (5 minutes)
6. Full meditation, which includes gently opening one's eyes and being mindful of the world of the moment, quietly attending, and waiting. When noticing something, be it a sight, sound, thought, or sensation, the individual must let it go and then resume attending, doing nothing else, and waiting for what comes next (5 minutes).

The experimental group received 30-minute individually administered, guided, chairside interventions during their hemodialysis sessions. This protocol has been found to be feasible and effective for patients undergoing hemodialysis [6]. Smith (2005) explained in his ABC relaxation theory that at least two and preferably five weekly 30-minute sessions of actual training of mind-body therapies should be provided to evoke relaxation, relieve stress, and improve health in general populations. However, for hemodialysis patients, it has been suggested that brief program formatting with at least 400 total minutes may lead to greater health benefits. Accordingly, the experimental group received 30-minute mindfulness meditation sessions 3 times a week for 5 weeks (450 minutes) The participants also received a 2-hour foundation course which was introduced and supervised by one of the study researchers prior to the actual training sessions and which taught the participants the intervention basics, benefits, protocol, and method of access. To ensure the consistent delivery of the intervention, the researcher recorded the intervention instructions in Arabic based on the intervention protocol and sent the audio-recorded instructions to the participants via WhatsApp or email. The audio-recorded intervention contents were validated by 2 psychologists and experts in meditation. The recorded intervention instructions were accessed by the participants during the sessions using their cell phones and headsets, as recommended. This method allowed for up to 3-5 participants to listen to the instructions and perform the intervention simultaneously.

The researcher who was responsible for developing the study intervention and supervising the intervention delivery was an experienced mind-body practitioner who had received a 4-day training course on mindfulness meditation. The researcher attended the sessions to manage any potential interruptions and evaluate the intervention delivery. The participants' privacy was maintained using curtains surrounding each participant during the intervention. The participants were asked not to share any information related to the intervention with the participants in the control group.

The participants in the control group were instructed to sit with their eyes closed and relaxed for 30 minutes 3 times a week for 5 weeks during hemodialysis sessions to control for the nonspecific effects of social interaction and environment. The timings of the control group sessions were similar to those of the experimental group, whereby if a given experimental group intervention lasted for 30 minutes, the control group participants would be asked to sit with their eyes closed and relax for 30 minutes also.

Procedure

First, the permission from the instruments used in the study was obtained. Recruitment of participants was conducted by one of the study researchers after obtaining approval to conduct the study from the hospital administrators. The study purposes and protocol were explained to the patients in detail. Patients who agreed to participate in the study and met the eligibility criteria were asked to sign a consent form, and the participating patients were then randomly assigned to the two study groups. The baseline measurements of the study variables were taken using the self-report questionnaires, which were administered by a research assistant who was not involved in any other parts of the study. The study variables were also measured two weeks post the start of the intervention and at the end of the final session for both groups under the same conditions. All measurements were privately taken at the dialysis center.

Data Analysis

SPSS version 25 was used to analyze the collected data. Prior to the main analysis, outliers and missing data were examined and managed as appropriate. Then, the assumptions of the statistical tests used, normality using histogram graph, homogeneity of variance, and sphericity were checked and managed as appropriate. Mauchly's test of sphericity is used to assess whether the sphericity assumption has been violated. When Mauchly's test of sphericity was significant (p < .05), the degrees of freedom were corrected using Greenhouse-Geisser estimates of sphericity. The comparability of the two groups was evaluated in terms of demographic characteristics and the baseline measurements of the dependent variables using t-test and Chi square, based on the measurements of the dependent variables. The main analysis was conducted with repeated-measures ANOVA (mixed design: within and between groups). A P-value of 0.0125 was set as the significance level for the main analysis tests. The p-value was adjusted due to multiple testing by dividing the p-value of .05 by 4 (number of dependent variables).

Ethical Considerations

The study proposal was approved by the Institutional Review Board at Jordan University of Science and Technology and the Kuwaiti Ministry of Health (Number of approval: 78/136/2020). The study was conducted in accordance with the Declaration of Helsinki. The participants were asked to sign informed consent forms which included an explanation of the study purpose and protocol, in addition to a statement indicating that the participants had the right to refuse to participate or withdraw from the study at any time without consequences. The participants were assured that their information would not be made available to others without their consent. The study data were stored in a locked locker after all names were replaced by numbers.

ELIGIBILITY:
Inclusion Criteria:

* being a patient with ESRD undergoing hemodialysis three times a week
* being aged 18 years old or over
* being able to read and write in Arabic.

Exclusion Criteria:

* being a patient with cognitive dysfunction or mental retardation
* taking psychopharmacological drugs
* undergoing psychotherapy
* practicing any type of relaxation techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Trait Mindfulness | 6 weeks
  An Arabic version of the Mindful Attention Awareness Scale (MAAS) was used to measure trait mindfulness. The MAAS is one-dimensional and comprises 15 items measured on a six-point Likert-type scale ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher scores indicating higher levels of trait mindfulness. The Arabic MAAS has been shown to have excellent internal consistency and convergent validity among an Arab population. In our study, the Chronbach's alpha values for the MAAS was 0.93.
Perceived stress | 6 weeks
  The Arabic version of the Perceived Stress Scale (PSS) was used to measure the degree to which situations in one's life are appraised as stressful (unpredictable, uncontrollable, or overloaded). The scale comprises 10 items which are measured on a 5-point Likert scale (0=never, 4= very often) and which are relatively free of content specific to any subpopulation group. The total possible score ranges from 0 to 40, with higher scores indicating higher levels of perceived stress (stress appraisal) [22]. The Arabic PSS has been shown to have adequate reliability and validity and is considered a suitable instrument for assessing perceived stress in Arab people [21]. In the current study, the Chronbach's alpha values for the PSS was 0.82.
Emotion regulation | 6 weeks
  The Arabic version of the Emotion Regulation Questionnaire (ERQ) was used to assess emotion regulation among the study sample. The questionnaire items are scored on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree) and are divided into two subscales, namely cognitive reappraisal and expressive suppression. Higher scores indicate greater emotion regulation abilities. The Arabic version of the ERQ has shown valid and reliable results among the Arab population. In our study, the Chronbach's alpha values for the ERQ was 0.81.
kidney disease-quality of life | 6 weeks
  The Arabic version of the Kidney Disease-Quality of Life questionnaire (KDQOL-36) is used to assess kidney disease-related quality of life and consists of four subscales: Generic Core [Physical Component Summary (PCS, 12 items) and Mental Component Summary (MCS, 12 items)]; Symptoms/Problems (12 items); Burden of Kidney Disease (4 items), and Effects of Kidney Disease (8 items). The scores of the different subscales are calculated according to the KDQOL-36 scoring system. Raw, pre-coded numeric values for each item are transformed linearly to a range of 0 to 100, with higher scores reflecting better kidney disease-quality of life. The Arabic version used in this study showed good psychometric qualities among Arab patients with chronic renal failure. In our study, the Chronbach's alpha values for KDQOL-36 was 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tohme F, Mor MK, Pena-Polanco J, Green JA, Fine MJ, Palevsky PM, Weisbord SD. Predictors and outcomes of non-adherence in patients receiving maintenance hemodialysis. Int Urol Nephrol. 2017 Aug;49(8):1471-1479. doi: 10.1007/s11255-017-1600-4. Epub 2017 Apr 28. PMID 28455663
- [Background] Kraus MA, Fluck RJ, Weinhandl ED, Kansal S, Copland M, Komenda P, Finkelstein FO. Intensive Hemodialysis and Health-Related Quality of Life. Am J Kidney Dis. 2016 Nov;68(5S1):S33-S42. doi: 10.1053/j.ajkd.2016.05.023. PMID 27772641
- [Background] Shariaty Z, Mahmoodi Shan GR, Farajollahi M, Amerian M, Behnam Pour N. The effects of probiotic supplement on hemoglobin in chronic renal failure patients under hemodialysis: A randomized clinical trial. J Res Med Sci. 2017 Jun 21;22:74. doi: 10.4103/jrms.JRMS_614_16. eCollection 2017. PMID 28717371
- [Background] Haramaki Y, Kabir RS, Abe K, Yoshitake T. Promoting Self-Regulatory Management of Chronic Pain Through Dohsa-hou: Single-Case Series of Low-Functioning Hemodialysis Patients. Front Psychol. 2019 Jun 20;10:1394. doi: 10.3389/fpsyg.2019.01394. eCollection 2019. PMID 31281283
- [Background] Thomas Z, Novak M, Platas SGT, Gautier M, Holgin AP, Fox R, Segal M, Looper KJ, Lipman M, Selchen S, Mucsi I, Herrmann N, Rej S. Brief Mindfulness Meditation for Depression and Anxiety Symptoms in Patients Undergoing Hemodialysis: A Pilot Feasibility Study. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2008-2015. doi: 10.2215/CJN.03900417. Epub 2017 Oct 12. PMID 29025788
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] Garland E, Gaylord S, Park J. The role of mindfulness in positive reappraisal. Explore (NY). 2009 Jan-Feb;5(1):37-44. doi: 10.1016/j.explore.2008.10.001. PMID 19114262
- [Background] Cho IH, Suh SR, Jang KH. Stress coping resources of hemodialysis patients: Mindfulness. International Journal of Advanced Nursing Education and Research. 2017;2(1):153-8
- [Background] Kabat-Zinn, Mindfulness-based interventions in context: past, present, and future, Clin. Psychol. Sci. Pract 2003;10(2):144-156
- [Background] Igarashi NS, Karam CH, Afonso RF, Carneiro FD, Lacerda SS, Santos BF, Kozasa EH, Rangel EB. The effects of a short-term meditation-based mindfulness protocol in patients receiving hemodialysis. Psychol Health Med. 2022 Jul;27(6):1286-1295. doi: 10.1080/13548506.2021.1871769. Epub 2021 Jan 15. PMID 33449820
- [Background] Adamoli AN, Razzera BN, Ranheiri MF, Colferai RN, Russell TA, Noto AR, et al. Mindfulness-Based Intervention Performed During Hemodialysis: an Experience Report. Trends in Psychology 2021;29(2):320-40
- [Background] Gross CR, Reilly-Spong M, Park T, Zhao R, Gurvich OV, Ibrahim HN. Telephone-adapted Mindfulness-based Stress Reduction (tMBSR) for patients awaiting kidney transplantation. Contemp Clin Trials. 2017 Jun;57:37-43. doi: 10.1016/j.cct.2017.03.014. Epub 2017 Mar 22. PMID 28342990
- [Background] Noorifard M, Neshat Doost H T, Sajjadian I. Comparative of Mindfulness with Memory Specificity Training (MEST) on Cognitive Emotion Regulation Strategies in Hemodialysis Patients. MEJDS 2019; 9:46-46
- [Background] Moosavi Nejad M, Shahgholian N, Samouei R. The effect of mindfulness program on general health of patients undergoing hemodialysis. J Educ Health Promot. 2018 Jun 12;7:74. doi: 10.4103/jehp.jehp_132_17. eCollection 2018. PMID 29963567
- [Background] Nassim M, Park H, Dikaios E, Potes A, Elbaz S, Mc Veigh C, Lipman M, Novak M, Trinh E, Alam A, Suri RS, Thomas Z, Torres-Platas S, Vasudev A, Sasi N, Gautier M, Mucsi I, Noble H, Rej S. Brief Mindfulness Intervention vs. Health Enhancement Program for Patients Undergoing Dialysis: A Randomized Controlled Trial. Healthcare (Basel). 2021 Jun 1;9(6):659. doi: 10.3390/healthcare9060659. PMID 34205915
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Rayan A, Ahmad M. The psychometric properties of the mindful attention awareness scale among Arab parents of children with autism spectrum disorder. Arch Psychiatr Nurs. 2018 Jun;32(3):444-448. doi: 10.1016/j.apnu.2018.01.001. Epub 2018 Jan 3. PMID 29784228
- [Background] Almadi T, Cathers I, Hamdan Mansour AM, Chow CM. An Arabic version of the perceived stress scale: translation and validation study. Int J Nurs Stud. 2012 Jan;49(1):84-9. doi: 10.1016/j.ijnurstu.2011.07.012. Epub 2011 Aug 17. PMID 21851941
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Keshky ME. Factor Structure, Reliability and Validity of the Arabic Version of the Emotion Regulation Questionnaire (ERQ) in a Sample of Saudi Children and Adolescents. Int J Psychol Behav Sci 2018;8(2):22-30
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Elamin S, E Elbasher AH, E Ali SE, Abu-Aisha H. Arabic translation, adaptation, and validation of the kidney disease quality of life short-form 36. Saudi J Kidney Dis Transpl. 2019 Nov-Dec;30(6):1322-1332. doi: 10.4103/1319-2442.275476. PMID 31929279
- [Background] Kalantar-Zadeh K, Unruh M. Health related quality of life in patients with chronic kidney disease. Int Urol Nephrol. 2005;37(2):367-78. doi: 10.1007/s11255-004-0012-4. PMID 16142573
- [Background] Smith JC. Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company; New York, NY, 2005 Mar 4.
- [Background] Murakami H, Katsunuma R, Oba K, Terasawa Y, Motomura Y, Mishima K, Moriguchi Y. Neural Networks for Mindfulness and Emotion Suppression. PLoS One. 2015 Jun 17;10(6):e0128005. doi: 10.1371/journal.pone.0128005. eCollection 2015. PMID 26083379
- [Background] Shafiee MA, Chamanian P, Shaker P, Shahideh Y, Broumand B. The Impact of Hemodialysis Frequency and Duration on Blood Pressure Management and Quality of Life in End-Stage Renal Disease Patients. Healthcare (Basel). 2017 Sep 2;5(3):52. doi: 10.3390/healthcare5030052. PMID 28869490
- [Derived] Alhawatmeh H, Alshammari S, Rababah JA. Effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in hemodialysis patients: A randomized controlled trial. Int J Nurs Sci. 2022 Mar 8;9(2):139-146. doi: 10.1016/j.ijnss.2022.03.004. eCollection 2022 Apr. PMID 35509694

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT05176730/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT05176730/ICF_001.pdf